CLINICAL TRIAL: NCT00800657
Title: Stem-Cells and Heart Failure in Several Ethiologies. Alternative Indication With Cardiac Resynchronization
Brief Title: Stem Cells and Resynchronization Cardiac
Acronym: RCT and SCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Molestias Cardiovasculares (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Oswaldo Tadeu Greco, IMC - Instituto de Moléstias Cardiovasculares
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HFRCTC1; HFRCTC1
Record Dates: First submitted 2008-11-12; First posted 2008-12-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization; Dilated Cardiomyopathy; Stem Cells Therapy; Heart Failure; Stem Cells/Cardiac Pacing, Artificial
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Pacing and Stem Cells Implantations. — Implantation of Cardiac Ressyncrhonization combined with the implantation of Stem Cells Hematopoietics.
Procedure: Pacing and Stem Cells Implantation — Pacing and Stem Cells Implantation.

SUMMARY:
Same patients with dilated myocardiopathies with large areas of fibrosis has not been as successful after Cardiac Resynchronization Therapy, for Heart Failure patients in functional class III or IV. Therefore the investigators have decided to associate the Stem-Cell implant with Cardiac Resynchronization Therapy in these patients.

DETAILED DESCRIPTION:
About 120cc of blood are collected from the iliac bone marrow under epidural anesthesia.In the cell therapy lab this blood is harvested and mononuclear cells are separated.This procedure takes roughly 4 hours.After dilution the mononuclear cells are injected into the cardiac muscles with fibroses area through 20 shots.This procedure is indicated for patients with cardiac ischemia and left ventricular dysfunction(desynchrony), on whom all the others known therapies have failed.

ELIGIBILITY:
* Dilated Cardiomyopathy
* Heart Failure
* Optimized Therapeutics
* Ventricular Desynchrony
* Functional Class III or IV
* Ejection Fraction(Echo/ Sympson) < 35%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction(EF)-(Eco- Sympson):It is the comparison of these measurements between late pre and post operative. NYHA: Comparison of these measurements between late pre and post operative. | 24 months

SECONDARY OUTCOMES:
Ejection Fraction (Echo/Sympson) and functional class(NYHA). | 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Oswaldo Tadeu Greco, PhD, Principal Investigator — IMC - Institute of Hearth Diseases; Oswaldo Tadeu Greco, PhD, Principal Investigator — IMC- Institute of Hearth Diseases
Locations (1):
- Imc - Instituto de Moléstias Cardiovasculares, São José do Rio Preto, São Paulo, Brazil

REFERENCES:
- [Result] Jacob JL, Salis FV, Ruiz MA, Greco OT. Labeled stem cells transplantation to the myocardium of a patient with Chagas' disease. Arq Bras Cardiol. 2007 Aug;89(2):e10-1. doi: 10.1590/s0066-782x2007001400014. English, Portuguese. PMID 17874006
- See also: Departamento de Estimulação Cardiaca e Arritmia. — http://deca.org.br